CLINICAL TRIAL: NCT00534573
Title: Comparison of Benzamide Derivates (Amisulpride, Moclobemide and Tiapride) as Treatment of Clozapine-induced Hypersalivation: Pilot Double Phase Study: Open and Double-blind
Brief Title: Benzamide Derivates as Treatment of Clozapine-induced Hypersalivation
Acronym: CIH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beersheva Mental Health Center (Other Government)
Collaborators: Tirat Carmel Mental Health Center (Other Government)
Responsible Party: Principal Investigator, Vladimir Lerner, A/Professor, Head of department, Beersheva Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LCK4569; ISRCTN4569; ISRCTN4569 (Other: ISRCTN4569)
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2009-11

CONDITIONS: Clozapine-induced Hypersalivation
MeSH Terms: interventions — Amisulpride; Moclobemide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moclobemide, (Active Comparator): treatment during 2 weeks
  Interventions: Drug: Amisulpride, Moclobemide
- Amisulpride (Active Comparator): Comparison
  Interventions: Drug: Amisulpride, Moclobemide

INTERVENTIONS:
Drug: Amisulpride, Moclobemide — Amisulpride 400 mg/d; Moclobemide 300 mg/d every medication for 2 week aith 2 week washout

SUMMARY:
Hypersalivation (sialorrhea or ptyalism) is known as a frequent, disturbing, uncomfortable adverse effect of clozapine therapy, and until now there is not enough effective treatment for this side effect leading to noncompliance.

In previous studies it was found that substitute benzamide derivatives with higher selective binding to the D2/D3 dopamine receptor - amisulpride and sulpiride may be effective in treatment of clozapine-induced hypersalivation (CIH). Today, in psychiatric practice in Israel, there are four medications which belong to substitute benzamide derivatives group: amisulpride, sulpiride, tiapride and moclobemide. We hypothesized that antisalivation effect is universal for the whole group of benzamide.

The aim of our study was to compare efficacy of amisulpride, moclobemide (reversible monoamine oxidase inhibitor-A (RIMAS)), and tiapride (dopamine D2 antagonist) as an additional possibility for management of CIH.

DETAILED DESCRIPTION:
The pilot study will be conducted in two mental health centers. In order to examine our hypothesis, we will use an add-on design. Into the study will be enrolled 50 patients with schizophrenia and schizoaffective disorder (males and females, 19-60 years old), according to the DSM-IV criteria, treated with clozapine and suffering from hypersalivation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years, male or female
* DSM-IV criteria for schizophrenia
* Clozapine treatment
* At least 2 scores on the Nocturnal Hypersalivation Rating Scale (NHRS)

Exclusion Criteria:

* Evidence of organic brain damage, mental retardation, alcohol or drug abuse

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2008-11; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Hypersalivation will be assessed by subjective and objective tools. Clinical global impression (CGI) patient's self assessment will be taken as subjective tool and NHRS as an objective assessment tool. | every two days
  NHRS, CGI

SECONDARY OUTCOMES:
CGI, NHRS | two weeks
  CGI, NHRS

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Lerner, MD, PhD, Principal Investigator — Be'er Sheva Mental Health Center; Anatoly Kreinin, MD, PhD, Principal Investigator — Tirat HaKarmel Mental Health Center; Chanoch Miodownik, MD, Study Director — Be'er Sheva Mental Health Center; Igor Libov, Study Director — Be'er Sheva Mental Health Center; Alexander Grinshpoon, MD, Study Director — Tirat HaKarmel Mental Health Center; Diana Shestakova, MD, Study Director — Tirat HaKarmel Mental Health Center
Locations (1):
- Be'er Sheva Mental Health Center, Tirat HaKarmel Mental Health Center, Be'er Sheva, Haifa, Israel

REFERENCES:
- [Derived] Kreinin A, Miodownik C, Sokolik S, Shestakova D, Libov I, Bergman J, Lerner V. Amisulpride versus moclobemide in treatment of clozapine-induced hypersalivation. World J Biol Psychiatry. 2011 Dec;12(8):620-6. doi: 10.3109/15622975.2010.527370. Epub 2010 Oct 21. PMID 20964499